CLINICAL TRIAL: NCT03838887
Title: Comparison Between Uterine Artery Doppler and Placental Vascular Indices in Prediction of Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Sherif Elsirgany, Researcher ,Family Planning and Reproductive Health Department, National Research Centre, Egypt
Other Study IDs: placental vascular indices
Record Dates: First submitted 2019-02-03; First posted 2019-02-12 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Pregnant women:
  1. Age between 18-35 years
  2. Parity: primigravidas and multiparas.
  3. Have no history of preeclampsia or eclampsia.
  4. Have no history of chronic hypertension.
  5. Not diabetic.
  6. Not have antiphospholipid syndrome.
  7. Not have autoimmune disease such as SLE
  Interventions: Device: ultrasound machine
- High risk group: Pregnant women with:
  1. History of preeclampsia -Eclapmsia
  2. Chronic hypertension
  3. Diabetic
  4. Antiphospholipid syndrome.
  5. Autoimmune syndrome such as SLE.
  Interventions: Device: ultrasound machine

INTERVENTIONS:
Device: ultrasound machine — Ultrasound machine with a vocal software

SUMMARY:
• Preeclampsia is a multisystem disorder that can cause considerable maternal and fetal morbidity and mortality. Late preeclampsia (with delivery >34 weeks) is more frequent and less serious than early preeclampsia (with delivery <34 weeks). Poor early placentation has been especially associated with early disease. Early identification of women at risk of preeclampsia is currently a crucial aim of antenatal care since they may benefit from prophylactic treatment and increased surveillance.

DETAILED DESCRIPTION:
* The introduction of three-dimensional (3D) ultrasound techniques, with the option of calculating placental volume and measuring vascular indices, has created an excellent opportunity to study early changes in the uteroplacental circulation space, which includes the maternal spiral arteries and the intervillous space. This technology may allow a more direct evaluation of the abnormal placentation process thought to herald the development of preeclampsia.
* The aim of this study was to assess the usefulness of placental volume and 3D vascular indices as reliable predictors of early preeclampsia in comparison to uterine artery Doppler

ELIGIBILITY:
Inclusion Criteria:

* A. Control group: Pregnant women:

  1. Age between 18-35 years
  2. Parity: primigravidas and multiparas.
  3. Have no history of preeclampsia or eclampsia.
  4. Have no history of chronic hypertension.
  5. Not diabetic.
  6. Not have antiphospholipid syndrome.
  7. Not have autoimmune disease such as SLE.

B. High risk group: Pregnant women with:

1. History of preeclampsia -Eclapmsia
2. Chronic hypertension
3. Diabetic
4. Antiphospholipid syndrome.
5. Autoimmune syndrome such as SLE.

Exclusion Criteria:

* • Smoking

  * Dichorionic placentae
  * Fetal anomaly
  * Uterine fibroid at the site of placental implantation
  * Subchorionic hematoma

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — examination of pregnant women
Study Population: All pregnant women will be examined for antenatal care in the outpatient clinic and fetal medicine unit of obstetrics and gynecology department then they will be divided into two groups control and high risk
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
placental vascular indices in prediction of preeclampsia | one year
  placental vascular indices in prediction of preeclampsia compared to uterine artery doppler in prediction of preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided